CLINICAL TRIAL: NCT05895890
Title: Study of the Evolution of the Intestinal Microbiome (Taxonomic and Functional Composition) During Alcoholic Liver Disease
Brief Title: French National MICMAF Cohort
Acronym: MICMAF
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 200312; 2019-A01331-56 (Other: French Agency for the Safety of Health Products)
Record Dates: First submitted 2023-02-20; First posted 2023-06-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Alcoholic Liver Disease
Keywords: Alcoholic; Liver Disease; Intestinal microbiome; Addiction; Depression
MeSH Terms: conditions — Liver Diseases, Alcoholic; Liver Diseases; Behavior, Addictive; Depression | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, saliva, serum and whole blood samples from research samples will be collected in a biological collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohorte: The study will include a population of patients with excessive alcohol consumption seen in consultation or hospitalized for alcohol addiction problems and/or exploration of alcohol-related liver damage
  Interventions: Genetic: Sequential sampling (stool, saliva, serum) .

INTERVENTIONS:
Genetic: Sequential sampling (stool, saliva, serum) . — Sequential sampling (stool, saliva, serum) prior to the occurrence of AAH episodes in heavy drinking patients to identify protective or deleterious profiles.

SUMMARY:
Excessive alcohol consumption is a major public health problem, particularly in France. It is the leading cause of cirrhosis and hepatocellular carcinoma. Among subjects with heavy alcohol consumption, the majority of patients develop fatty liver overload (steatosis), but only 10 to 35% develop acute alcoholic hepatitis (AAH) and 8 to 20% progress to cirrhosis. Steatosis is the earliest lesion, rapidly reversible after abstinence from alcohol. On the other hand, the occurrence of AAH leads to a strong progression of fibrosis. The investigators have shown on serial liver biopsies that a subgroup of heavy drinkers develop episodes of AAH and progress to cirrhosis. Therefore, factors other than the amount of alcohol consumed alone influence the development and progression of alcoholic liver disease (ALD). Among these factors, it is now accepted that the gut microbiome plays an important role in the pathogenesis of ALD. Increased intestinal permeability and activation of the innate immune system by lipolysaccharide (LPS) of digestive origin is a key factor in the initiation of AAH. The alteration of the intestinal barrier induced by alcohol abuse seems to involve dysbiosis. Furthermore, the investigatorshave shown that the sensitivity of the liver to alcohol toxicity is transmissible from humans to mice via the gut microbiome. Despite these advances, the causal relationship between mycobiome disruption and ALD in humans requires confirmation in prospective studies.

The intestinal microbiome represents all the microorganisms found in the digestive tract: bacteria (bacterial microbiome), viruses (virome), fungi (mycobiome).

Recent data point to the role of disturbances of the mycobiome and the virome in human pathology. The intestinal virome consists of two major types of viruses: eukaryotic RNA and DNA viruses that infect host cells and prokaryotic or bacteriophage viruses that infect the bacterial microbiome. Recent evidence suggests that the virome participates in immune system homeostasis. Infection of axenic mice with murine norovirus restores the functionality of intestinal lymphocytes. However, the involvement of the intestinal virome in ALD has never been studied.

Cessation of alcohol consumption has a beneficial effect in all stages of ALD . It reduces the risk of complications of cirrhosis and, for early stages of liver damage, prevents progression to advanced stages (severe AAH and cirrhosis). Unfortunately, most patients with alcohol addiction do not achieve long-term abstinence or significant reduction in their consumption despite psychological and medical support. Depression and anxiety are also associated with gut dysbiosis in humans. The causal role, at least partial, of this dysbiosis in addictive phenomena, whether alcohol or other addictions such as cocaine, has been shown. Thus, the modification of MI influences the addictive behavior of cocaine-dependent mice (. All these data show the major role of the microbiota-central nervous system (CNS) axis in mental disorders such as alcohol addiction and its consequences (craving, depression, anxiety). This interaction is mediated by several mechanisms such as the production of active metabolites by the intestinal microbiome and the translocation of bacteria or bacterial derivatives.

Primary Objective:

To characterize temporal changes in the gut microbiome (bacterial, viral, and fungal) within sequential specimens (stool, saliva, serum) prior to the occurrence of acute alcoholic hepatitis episodes

Secondary Objectives:

* Demonstrate that specific fecal, serum, or saliva microbiome profiles (bacterial, viral, and fungal) can predict the progression of alcoholic liver disease to severe alcoholic hepatitis, fibrosis, and cirrhosis.
* Characterize changes in the composition of the gut microbiome (bacterial, viral and fungal) associated with the progression of alcoholic liver disease to severe alcoholic hepatitis and cirrhosis.
* Characterize the changes in the microbiome during alcohol withdrawal.
* Identify microbiome profiles associated with alcohol dependence and anxiety-depressive events related to alcohol addiction.
* To identify bacterial species with a protective effect in alcoholic liver disease.
* To identify beneficial bacterial species against alcohol dependence.
* To study the microbiome-host interaction in alcoholic liver disease and alcohol addiction.
* To identify microbiome profiles with prognostic value in severe alcoholic hepatitis and alcoholic cirrhosis.

Number of centers: 7 Number of subjects expected 1000 Population concerned: The study will include a population of patients with excessive alcohol consumption seen in consultation or hospitalized for alcohol addiction problems and/or exploration of alcohol-related liver damage Inclusion period: January 2020 - January 2030 Patient observation period: 5 to 20 years Study duration: 30 years

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Average alcohol consumption of more than 20 g per day in women and 30 g per day in men during the previous year;
* Patients seen in consultation or hospitalized for assessment of alcoholic liver disease and management of alcohol addiction;
* Having given their consent to participate in this study;
* Affiliated to a social security system (beneficiary or beneficiary's right).

Exclusion Criteria:

* Antibiotic, probiotic or prebiotic treatment within the previous 3 months ;
* Digestive hemorrhage, acute pancreatitis, acute or chronic diarrhea (except diarrhea related to excessive alcohol consumption) or chronic inflammatory bowel disease;
* Another cause of liver damage;
* A serious associated pathology (respiratory failure, heart failure, severe psychiatric disorders, active cancer).
* Patient under guardianship or curatorship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include a population of patients with excessive alcohol consumption seen in consultation or hospitalized for alcohol addiction problems and/or exploration of alcohol-related liver damage.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2043-02-01 (Estimated); Study Completion 2053-02-01 (Estimated)

PRIMARY OUTCOMES:
Temporal changes in the gut microbiome | every 6 months until 240 months
  Differences in gut microbiome composition between inclusion and different follow-up visits

SECONDARY OUTCOMES:
Differences in gut microbiome composition as a function of the rate of progression of liver fibrosis | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique, the rate of progression of liver fibrosis, as measured by median elasticity (kPa/year)
Differences in gut microbiome composition at inclusion between patients with and without the development of severe acute alcoholic hepatitis or cirrhosis between inclusion and different follow-up visits. | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique
Differences in gut microbiome composition at baseline between failed and weaned patients and between baseline and follow-up visits. | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique,
Differences in gut microbiome composition as a function of craving intensity, depression and anxiety. | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique
The correlation between gut microbiome, host genotype and FAD severity. | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique
Effect of bacteria identified as beneficial, on mouse models of alcoholic liver disease, depression and anxiety. | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique
The association between the gut microbiome and the prognosis of patients with acute alcoholic hepatitis or cirrhosis. | every 6 months until 240 months
  Differences in the composition of the gut microbiome, analyzed using the metagenomic technique

CONTACTS AND LOCATIONS:
Overall Officials: Cosmin Voican, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cosmin Voican, Clamart, Île-de-France Region, France